CLINICAL TRIAL: NCT04285060
Title: Safety and Efficacy on Functional Mobility Following Samsung GEMS-H Device Training in Sub-Acute and Chronic Stroke: A Pivotal Study
Brief Title: Safety and Efficacy of Samsung GEMS-H Device Training in Sub-Acute and Chronic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Electronics (Industry)
Collaborators: Shirley Ryan AbilityLab (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 00210372
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Stroke; Chronic Stroke
Keywords: Stroke; Exoskeleton
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Training Group (Experimental): All participants are assigned to the training group with the Samsung GEMS-H.
  Interventions: Device: Samsung GEMS-H

INTERVENTIONS:
Device: Samsung GEMS-H — Subjects will participate in 18 sessions of training in the outpatient clinic with a licensed physical therapist. Therapy sessions will include 30 minutes of task specific training and another 15 minutes of the session can be used to focus on patient specific goal areas related to functional mobility and balance. Training sessions will occur 2-3 times a week for 6-8 weeks to complete the training protocol.

SUMMARY:
A single-site, interventional, single-arm trial to evaluate the safety and efficacy on functional mobility following Samsung GEMS-H (Gait Enhancing and Motivating System - Hip) device training in participants with sub-acute and chronic stroke.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 30-days post stroke
* Age: 18-85 Years
* Initial gait speed of ≥ 0.4 m/s and ≤ 0.8 m/s
* Adequate cognitive function (MMSE score >17)
* Ability to walk at least 10m with maximum 1 person assist
* Physician approval for patient participation
* Able to safely fit into device specifications and tolerate minimum assistance

Exclusion Criteria:

* ≤90 days post major orthopedic surgery (i.e. hip, knee, and/or ankle joint replacement)
* ≤ 6 months post coronary artery bypass graft (CABG) or cardiac valve procedure
* Severe osteoporosis as indicated by physician medical clearance
* Serious cardiac conditions (hospitalization for myocardial infarction or heart surgery within 3 months, history of congestive heart failure, documented serious and unstable cardiac arrhythmias, hypertrophic cardiomyopathy, severe aortic stenosis, angina or dyspnea at rest or during activities of daily living)
* Pregnancy
* Uncontrolled hypertension
* Lower extremity fracture
* Modified Ashworth Spasticity ≥3 in hip flexor or extensor
* Preexisting neurological disorders such as Parkinson's disease, Amyotrophic Lateral Sclerosis (ALS), Multiple Sclerosis (MS), dementia
* History of: major head trauma, lower extremity amputation, non-healing ulcers of a lower extremity, ongoing active infections, legal blindness, or a history of significant psychiatric illness
* Participating in any other structured outpatient, home health physical therapy program, or another clinical trial that according to the Principal Investigator is likely to affect study outcome or confound results.

TMS-Specific Exclusion Criteria

* Pacemakers, metal implants in the head region
* History of unexplained, recurring headaches, epilepsy/seizures/skull fractures or skull deficits
* Medications that lower seizure threshold
* History of concussion in last 6 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-02-12 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of device related adverse events | Duration of study participation (estimated 6 months)
  Safety will be assessed by the number of device related adverse events throughout the duration of the study
10 Meter Walk Test (Self-selected walking speed) (10MWT-SS) | Baseline, Post-Intervention (estimated 8 weeks)
  Change in self-selected walking speed measured without the device

SECONDARY OUTCOMES:
6 Minute Walk Test (6MWT) | Baseline, Post-Intervention (estimated 8 weeks)
  Change in walking endurance measured without the device
Berg Balance Scale (BBS) | Baseline, Post-Intervention (estimated 8 weeks)
  Changes in functional balance measured without the device
Functional Gait Assessment (FGA) | Baseline, Post-Intervention (estimated 8 weeks)
  Change in functional balance measured without the device

OTHER OUTCOMES:
Incidence of device malfunctions | Duration of study (estimated 12 months)
  Device reliability will be assessed by the number of device malfunctions throughout the duration of the study
ActiGraph activity monitor | Duration of study participation (estimated 4 months)
  Changes in average daily step count
Transcranial Magnetic Stimulation (TMS) | Baseline, Post-Intervention (estimated 8 weeks)
  Measure changes in descending corticospinal drive to the lower limb muscles
10 Meter Walk Test (Self-selected walking speed) (10MWT-SS) | Baseline, Mid-Intervention (estimated 4 weeks), 1 month Post-Intervention (1 month follow-up)
  Changes in self-selected walking speed measured without the device
10 Meter Walk Test (Fastest walking speed) (10MWT-FS) | Baseline, Mid-Intervention (estimated 4 weeks), Post-Intervention (estimated 8 weeks), 1 month Post-Intervention (1 month follow-up)
  Changes in fastest walking speed measured without the device
10 Meter Walk Test (Self-selected walking speed) (10MWT-SS) with the device | Baseline, Mid-Intervention (estimated 4 weeks), Post-Intervention (estimated 8 weeks), 1 month Post-Intervention (1 month follow-up)
  Changes in self-selected walking speeds between two conditions (with and without the device)
10 Meter Walk Test (Fastest walking speed) (10MWT-FS) with the device | Baseline, Mid-Intervention (estimated 4 weeks), Post-Intervention (estimated 8 weeks), 1 month Post-Intervention (1 month follow-up)
  Changes in fastest walking speeds between two conditions (with and without the device)
6 Minute Walk Test (6MWT) | Baseline, Mid-Intervention (estimated 4 weeks), 1 month Post-Intervention (1 month follow-up)
  Changes in walking endurance measured without the device
6 Minute Walk Test (6MWT) with the device | Baseline, Mid-Intervention (estimated 4 weeks), Post-Intervention (estimated 8 weeks), 1 month Post-Intervention (1 month follow-up)
  Changes in walking endurance between two conditions (with and without the device)
Berg Balance Scale (BBS) | Baseline, Mid-Intervention (estimated 4 weeks), 1 month Post-Intervention (1 month follow-up)
  Changes in functional balance measured without the device
Functional Gait Assessment (FGA) | Baseline, Mid-Intervention (estimated 4 weeks), 1 month Post-Intervention (1 month follow-up)
  Change in functional balance measured without the device
5 Times Sit to Stand Test (5xSST) | Baseline, Mid-Intervention (estimated 4 weeks), Post-Intervention (estimated 8 weeks), 1 month Post-Intervention (1 month follow-up)
  Change in lower extremity strength measured without the device
Gait analysis using a gait mat | Baseline, Mid-Intervention (estimated 4 weeks), Post-Intervention (estimated 8 weeks), 1 month Post-Intervention (1 month follow-up)
  Changes in spatiotemporal parameters measured without the device
Fugl-Meyer Assessment of Motor Recovery after Stroke (FMA) | Baseline, Mid-Intervention (estimated 4 weeks), Post-Intervention (estimated 8 weeks), 1 month Post-Intervention (1 month follow-up)
  Changes in motor recovery measured without the device
Manual Muscle Testing (MMT) | Baseline, Post-Intervention (estimated 8 weeks), 1 month Post-Intervention (1 month follow-up)
  Changes in leg strength measured without the device
Modified Ashworth Test (MAS) | Baseline, Post-Intervention (estimated 8 weeks), 1 month Post-Intervention (1 month follow-up)
  Changes in leg spasticity measured without the device
Passive Range of Motion (PROM) | Baseline, Post-Intervention (estimated 8 weeks), 1 month Post-Intervention (1 month follow-up)
  Changes in passive range of motion in leg joints measured without the device
Modified Falls Efficacy Scale (mFES) | Baseline, Mid-Intervention (estimated 4 weeks), Post-Intervention (estimated 8 weeks), 1 month Post-Intervention (1 month follow-up)
  Changes in perception of balance and stability
Activities-specific and Balance Confidence Scale (ABC) | Baseline, Mid-Intervention (estimated 4 weeks), Post-Intervention (estimated 8 weeks), 1 month Post-Intervention (1 month follow-up)
  Changes in confidence in performing various ambulatory activities without falling
Stoke Impact Scale (SIS) | Baseline, Mid-Intervention (estimated 4 weeks), Post-Intervention (estimated 8 weeks), 1 month Post-Intervention (1 month follow-up)
  Changes in the measure of the impact of stroke on overall physical and cognitive function
Patient Health Questionnaire-9 (PHQ-9) | Baseline, Mid-Intervention (estimated 4 weeks), Post-Intervention (estimated 8 weeks), 1 month Post-Intervention (1 month follow-up)
  Changes in depression
Stroke Specific Quality of Life (SSQoL) | Baseline, Mid-Intervention (estimated 4 weeks), Post-Intervention (estimated 8 weeks), 1 month Post-Intervention (1 month follow-up)
  Changes in the health-related quality of life
Oxygen Consumption using Cosmed K4b2 | Baseline, Mid-Intervention (estimated 4 weeks), Post-Intervention (estimated 8 weeks), 1 month Post-Intervention (1 month follow-up)
  Changes in metabolic energy expenditure

CONTACTS AND LOCATIONS:
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Macaluso R, Giffhorn M, Prokup S, Cleland B, Lee J, Lim B, Lee M, Lee HJ, Madhavan S, Jayaraman A. Safety & efficacy of a robotic hip exoskeleton on outpatient stroke rehabilitation. J Neuroeng Rehabil. 2024 Jul 30;21(1):127. doi: 10.1186/s12984-024-01421-x. PMID 39080666